CLINICAL TRIAL: NCT07403279
Title: Effects of Sustained Natural Apophyseal Glides With and Without Integrated Neuromuscular Inhibition Technique on Pain, Range of Motion, and Function in Patients With Chronic Mechanical Neck Pain
Brief Title: Sustained Natural Apophyseal Glides With and Without Integrated Neuromuscular Inhibition Technique in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0175
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: Integrated Neuromuscular Inhibition Technique; Neck pain; Range of Motion; Sustained Natural Apophyseal Glides; Trigger points
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sustained Natural Apophyseal Glides With Integrated Neuromuscular Inhibition Technique (Experimental)
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Integrated Neuromuscular Inhibition Technique; Other: Standardized Physiotherapy Treatment
- Sustained Natural Apophyseal Glides (Active Comparator)
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Standardized Physiotherapy Treatment

INTERVENTIONS:
Other: Sustained Natural Apophyseal Glides — SNAGs were applied in three sets, with repetitions progressively increased from 6 to 10 over a period of four weeks, administered three times per week.
Other: Integrated Neuromuscular Inhibition Technique — The integrated neuromuscular inhibition technique comprised three steps: ischemic compression, strain-counterstrain technique, and muscle energy technique. The technique was applied to the upper trapezius, levator scapulae, sternocleidomastoid, and splenius capitis muscles. Muscle selection was based on palpatory examination performed prior to each treatment session. Each treatment session lasted 10 minutes, during which all three steps were repeated three times within a single session. The intervention was delivered three times per week for four weeks, resulting in a total of 12 treatment sessions.
  Arms: Sustained Natural Apophyseal Glides With Integrated Neuromuscular Inhibition Technique
Other: Standardized Physiotherapy Treatment — Standardized physiotherapy included the application of an electrical hot pack at moderate intensity for 10 minutes. Transcutaneous electrical nerve stimulation (TENS) delivered in continuous mode at a frequency of 100 Hz for 15 minutes. Passive stretching was performed for cervical muscles prone to tightness, including the levator scapulae, sternocleidomastoid, upper trapezius, and scalene muscles, with a 30-second hold, three sets of ten repetitions, and a one-minute rest between sets. Scapular stabilization exercises, comprising shoulder shrugging and scapular retraction, were performed for 15 repetitions with a 6-second hold. Neck isometric exercises were repeated ten times with a 6-second hold. Cervical stabilization exercises were performed in two sets of ten repetitions per session, with each repetition held for ten seconds, a forty-second rest between repetitions, and a two-minute rest between sets.

SUMMARY:
The study was conducted to determine the effects of Sustained Natural Apophysial Glide with and without Integrated Neuromuscular Inhibition Technique on pain, range of motion and function in patients with chronic mechanical neck pain

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 18 to 45 years and both genders.
* Patient having neck-pain symptoms for more than 3 months duration.
* Spurling test, distraction test, upper limb tension test and shoulder abduction test negative upon assessment.
* The participants should have MTrPs in any one of these following cervical muscles which include levator scapulae, upper trapezius, splenius capitis and sternocleidomastoid muscles which may be active or latent.
* A score greater than twenty percent on NDI.
* Jump Sign when pressure is applied.
* Positive Simons criteria which contains following these 5 characteristics :(1) Pain on palpation (2) pain that is radiating (3) Tightened cord like structure in muscle fiber that is detectable upon palpation(4) Reduced Flexibility of that muscle (5) 'twitching response' on needling.
* Participants who described pain which is felt between spinous process of 1st thoracic vertebrae and superior nuchal line in posterior or posterolateral part of neck

Exclusion Criteria:

* Recent fracture, trauma (whiplash injury) and surgery in and around the shoulder and neck
* Neural disorders due to prolapsed intervertebral disc
* Carcinoma, Heart diseases, Metabolic disease in bone and joints
* Patients having history of osteoporosis, prolong steroid and analgesics use
* Unstable spine and open sores, Localized infection in neck
* Vertebrobasilar insufficiency.
* Cervical radiculopathy and myelopathy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to end of treatment at 4th weeks
  Numeric Pain Rating Scale is utilized to evaluate pain.This is a scale between 0 and 10 where 0 denotes no pain and 10 denotes the worst pain whereas 1-3 denotes mild pain 4-6 denotes moderate pain and 7-10 denotes severe pain.

SECONDARY OUTCOMES:
Neck Disability Index | From enrollment to the end of treatment at 4th weeks
  The Neck Disability Index is a self-reported questionnaire used to assess neck-related functional disability. It consists of 10 items addressing pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored on a 6-point scale (0-5), with a total score ranging from 0 to 50, where higher scores indicate greater disability. Scores are categorized as no disability (0-4), mild disability (5-14), moderate disability (15-24), severe disability (25-34), and complete disability (≥35).
Range of Motion Cervical Spine (Flexion) | From enrollment to the end of treatment at 4th week.
  Changes in cervical spine flexion range of motion at baseline and 4th week of intervention was measured using goniometer
Range of Motion Cervical Spine (Extension) | From enrollment to the end of treatment at 4th week
  Changes in cervical spine extension range of motion at baseline and 4th week of intervention was measured using goniometer.
Range of Motion Cervical Spine (Lateral Flexion) Right Side | From enrollment to the end of treatment at 4th week
  Changes in cervical spine lateral flexion on right side range of motion at baseline and 4th week of intervention was measured using goniometer.
Range of Motion Cervical Spine (Lateral Flexion) Left Side | From enrollment to the end of treatment at 4th week
  Changes in cervical spine lateral flexion on left side range of motion at baseline and 4th week of intervention was measured using goniometer.
Range of Motion Cervical Spine (Rotation) Right Side | From enrollment to the end of treatment at 4th week
  Changes in cervical spine rotation on right side range of motion at baseline and 4th week of intervention was measured using goniometer
Range of Motion Cervical Spine (Rotation) Left Side | From enrollment to the end of treatment at 4th week
  Changes in cervical spine rotation on left side range of motion at baseline and 4th week of intervention was measured using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Ph.D, Principal Investigator — Riphah International Universirty
Locations (1):
- Lahore General Hospital,Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd El-Azeim A, Grase M. Efficacy of Mulligan on electromyography activation of cervical muscles in mechanical neck pain: randomised experimental trial. Physiotherapy Quarterly. 2023;31(4):7-14.
- [Background] Shelke A, B AP, M GB, Kumaran SD, G PR. Immediate effect of craniocervical flexion exercise and Mulligan mobilisation in patients with mechanical neck pain - A randomised clinical trial. Hong Kong Physiother J. 2023 Dec;43(2):137-147. doi: 10.1142/S1013702523500154. Epub 2023 Jun 21. PMID 37583921
- [Background] Ali Ismail AM, Abd El-Azeim AS, El-Sayed Felaya EE. Integrated neuromuscular inhibition technique versus spray and stretch technique in neck pain patients with upper trapezius trigger points: a randomized clinical trial. J Man Manip Ther. 2024 Apr;32(2):141-149. doi: 10.1080/10669817.2023.2192899. Epub 2023 Mar 23. PMID 36951194
- [Background] Lytras DE, Sykaras EI, Christoulas KI, Myrogiannis IS, Kellis E. Effects of Exercise and an Integrated Neuromuscular Inhibition Technique Program in the Management of Chronic Mechanical Neck Pain: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2020 Feb;43(2):100-113. doi: 10.1016/j.jmpt.2019.03.011. Epub 2020 May 30. PMID 32482433
- [Background] Ozlu O, Sahin M. The effect of mulligan mobilization technique application in addition to conventional physiotherapy on pain and joint range of motion in people with neck pain. J Bodyw Mov Ther. 2024 Jul;39:225-230. doi: 10.1016/j.jbmt.2024.02.009. Epub 2024 Mar 5. PMID 38876630
- [Background] Ferdinand R, Kohilavani S. TO COMPARE THE EFFECTIVENESS OF INTEGRATED NEUROMUSCULAR INHIBITION TECHNIQUE VERSUS BOWEN TECHNIQUE ON UPPER TRAPEZIUS TRIGGER POINT IN SUBJECTS WITH MECHANICAL NECK PAIN
- [Background] Dhami H, Kaur J, Kaur M. Comparison of Integrated Neuromuscular Inhibition Technique versus Myofascial Release of Upper Trapezius on Neck Range of Motion and Dysfunction in Individuals with Nonspecific Neck Pain. Indian Journal of Physiotherapy & Occupational Therapy. 2022;16(4).
- [Background] Abhilash P. Comparison between immediate effect of integrated neuromuscular inhibition technique and active release technique on chronic neck pain and upper trapezius trigger points. 2024.
- [Background] Thakur R, Mande P, Lokwani M. Effectiveness of Integrated Neuromuscular Inhibition Technique and Instrument Assisted Soft Tissue Mobilisation in the Management of Upper Trapezius Myofascial Trigger Points. Indian Journal of Physiotherapy & Occupational Therapy. 2022;16(4).
- [Background] Shaukat S, Kiran Q, Hanif A, Saleem I, Paracha MS, Batool T. Role of Integrated Neuromuscular Inhibition Technique in Managing Upper Trapezius Trigger Points in Non-Specific Neck Pain: A Randomized Controlled Trial. Journal of Health, Wellness, and Community Research. 2025:e51-e.
- [Background] Tank KD, Choksi P, Makwana P. To study the effect of muscle energy technique versus mulligan snags on pain, range of motion and functional disability for individuals with mechanical neck pain: a comparative study. Int J Physiother Res. 2018;6(1):2582-87.
- [Background] Kocaman H, Yıldız NT, Canlı M, Alkan H. COMPARISON OF THE EFFECTS OF MULLIGAN MOBILIZATION TECHNIQUE COMBINED WITH CERVICAL STABILIZATION EXERCISES WITH THE EFFECTS OF CERVICAL STABILIZATION EXERCISES ALONE IN CHRONIC NECK PAIN: RANDOMIZED CONTROLLED STUDY. Karya Journal of Health Science. 2023;4(3):227-34.
- [Background] Malik SZ, Haider R, Razzaq A, Rehman AU, Zahra S. Comparison of MET and Mulligan Mobilization Snags in Reducing Neck Pain and Improving Functional Activities in Chronic Mechanical Neck Pain Patients. Journal of Health, Wellness and Community Research. 2025:e567-e.
- [Background] Naz S, Jamali N, Iftikhar A, Nawaz H, Iqbal T, Ghafoor F. Compare the Effectiveness of Mulligan (Nags & Snags) and McKenzie (Self-Stretching) On Improving the Pain and Functional Ability in Patient with Chronic Neck Pain: Effectiveness of Mulligan and McKenzie in Patient with Chronic Neck Pain. Pakistan Journal of Health Sciences. 2023:47-52